CLINICAL TRIAL: NCT05328427
Title: Discontinuation of Antiviral Therapy as a Strategy to Cure Hepatitis B
Acronym: STOP-B
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: Sahlgrenska University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STOP-B
Record Dates: First submitted 2022-03-25; First posted 2022-04-14 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Tin Fluorides

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stopping (Active Comparator): Discontinuation of nucleoside analogue treatment
  Interventions: Other: Stopping
- Continue (No Intervention): Treatment with nucleoside analogue continued

INTERVENTIONS:
Other: Stopping — Discontinuation of nucleoside analogue
  Arms: Stopping

SUMMARY:
Cirrhosis or cancer of the liver caused by hepatitis B virus (HBV) are major global health problems. Chronic HBV infection has become more common in Sweden with immigration. The risk of cancer and the availability of effective antivirals has led to more and more people receiving long-term treatment with antiviral drugs. The disadvantages of this treatment are that it does not have a defined duration and that it very rarely leads to the cure. Several published studies suggest that a large proportion of patients who discontinue antiviral therapy after at least three years may achieve lasting cure of the infection or at least do not need to resume treatment. The mechanism of this effect is not known, but it is thought to be due to the fact that the immune response, which is activated when the amount of virus increases after the end of treatment, becomes more effective in eradicating infected liver cells than it was before starting treatment. As a consequence of these findings updated guidelines for treatment of hepatitis B state that for patients that have received nucleoside analogue treatment for > 3 years, discontinuation is an accepted therapeutic alternative.

The purpose of the planned study is to investigate the results of discontinued treatment, in terms of clinical outcome as well as immunological and virological mechanisms. The aim is to include 120 patients at four regional infectious diseases clinics (in Gothenburg, Borås, Skövde and Trollhättan), of which 90 will be randomized to discontinue and 30 to continue antiviral treatment. Blood samples will be taken regularly to monitor the outcome and for detailed studies of viral antigens and nucleic acid in the blood and for specific analyzes of the cells of the immune system. The goal is to understand why the discontinued treatment in some patients activates an effective immune response and how such an effect can be predicted even before or early after the treatment is stopped.

ELIGIBILITY:
Inclusion Criteria:

* Nucleoside analogue treatment for HBeAg-negative chronic hepatitis B for at least 36 months.

Exclusion Criteria:

* Liver cirrhosis or liver cancer.
* Co-infection with HCV, HDV or HIV.
* Inability to understand study information and give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
HBsAg seronegativisation | 1 year
  Serum HBsAg becoming negative
HBsAg seronegativisation | 2 years
  Serum HBsAg becoming negative
HBsAg reduction | 1 year
  HBsAg reduction by > 1 log IU/mL
HBsAg reduction | 2 years
  HBsAg reduction by > 1 log IU/mL
Clinical responder | 2 years
  Sustained HBV DNA < 2000 IU/mL and normal ALT

SECONDARY OUTCOMES:
HBV-specific T cell activation | After 16 weeks
  Activation of HBV-specific T-cell responses, induced by incubating whole blood with HBV-core and HBsAg derived peptides for 48 hours, and investigated by measuring gamma interferon, chemokine and cytokine levels in plasma after centrifugation of the stimulated whole blood.

CONTACTS AND LOCATIONS:
Locations (1):
- Infectious Diseases Clinic, Sahlgrenska University Hospital, Gothenburg, VGR, Sweden

IPD SHARING:
Plan to Share IPD: No